CLINICAL TRIAL: NCT07284966
Title: Evaluation of Wear Comfort and Vision With Total 30 Multifocal Lenses Over 16 Hours of Wear
Brief Title: Comfort and Vision With TOTAL30 Multifocal Lenses
Status: Recruiting | Type: Observational
Sponsor: Scripps Poway Eyecare and Optometry (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor
Other Study IDs: JM-25-02
Record Dates: First submitted 2025-11-21; First posted 2025-12-16 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Myopia; Presbyopia; Astigmatism
MeSH Terms: conditions — Myopia; Presbyopia; Astigmatism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: TOTAL30 Multifocal — TOTAL30 Multifocal

SUMMARY:
This study is a single-arm, prospective, observational study conducted at one site to evaluate the comfort and vision of the TOTAL30 Multifocal (T30MF) contact lenses over the course of long wear days. The study will assess the proportion of positive subjective Visual Analog Scale (VAS) assessments of comfort and vision at 10, 12, 14, and 16 hours of wear on Days 1, 7, 14, and 30. Additionally, the study will explore subjective assessments of lens comfort using the CLDEQ-8 survey and measure logMAR visual acuity at both distance and near at Visit 1, Visit 2, and after 1 month of lens wear. Participants will undergo three site visits, with at-home surveys conducted at specified intervals to gather real-time data on comfort and vision.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible for the study if they meet the following criteria:

* Subjects who currently wear soft multi-focal contact lenses and score <12 on an entering CLDEQ-8 survey.
* Subjects who are >= 40 years old.
* Subjects who can and are willing to wear their lenses for 13 hours per day during the study period, and 16 hours per day when questionnaires are being taken.
* Willing to insert their contact lenses between 6:00 am and 8:00 am on the days when questionnaires will be taken.
* Vision correctable in soft multi-focal contact lenses to 20/25 (0.10 log MAR) or better in each eye at 6M.
* Must be able to be successfully fit into the prescription parameters available for Total30 MF contact lenses.
* Required to have a smartphone and receive push notifications.
* Willing to attend all study visits.
* Willing to be diligent about answering the timed surveys in a prompt manner.

Exclusion Criteria:

If any of the following exclusion criteria are applicable, the subject should not be enrolled in the study.

* Ocular anterior segment infection, inflammation, abnormality, or active disease that would contraindicate contact lens wear.
* Use of systemic or ocular medications for which contact lens wear could be contraindicated as determined by the investigator.
* Use of isotretinoin-derivatives.
* Use of lubricating drops.
* Monocular patients or patients fit with only 1 multifocal lens.
* Prior refractive surgery.
* History of herpetic keratitis, ocular surgery, or irregular cornea.
* Pregnant or lactating.
* Having participated in a clinical trial in the past 30 days.
* High-ADD habitual wearers using a different fitting approach than Alcon's multifocal fitting guide (e.g., J&J or CooperVision's fitting guide adopting a modified monovision approach).
* Are past rigid CL wearers.
* Have a history of being diagnosed with dry eye or ocular allergies.
* Have history of severe ocular trauma.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 40 years or older who currently wear soft multi-focal contact lenses.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2026-02-05 (Actual); Primary Completion 2027-01-21 (Estimated); Study Completion 2027-01-21 (Estimated)

PRIMARY OUTCOMES:
Patient-reported comfort level of the TOTAL30 Multifocal Lens | 16 hours of wear on specified days over a 30-day period
  Comfort level assessed using real-time patient-reported data collected at multiple time points throughout the day, with a focus on the end of the wear period. Patients are asked "What is your impression of the COMFORT of these study lenses?" and provide and answer from -50 (Extremely uncomfortable) to +50 (Extremely comfortable) using a sliding digital scale.

SECONDARY OUTCOMES:
Patient-reported vision quality with the TOTAL30 Multifocal Lens | 16 hours of wear on specified days over a 30-day period
  Vision quality assessed using real-time patient-reported data collected at various time points during the day. Patients are asked "What is your impression of the VISION quality of these study lenses?" and provide and answer from -50 (Poor quality) to +50 (Excellent quality) using a sliding digital scale.

OTHER OUTCOMES:
Contact Lens Dry Eye Questionnaire (CLDEQ-8) | After 1 month of wear
  A series of 8 questions that ask participants to rate eye discomfort, eye dryness, and blurry vision on a frequency scale (0 Never, 1 Rarely, 2 Sometimes, 3 Frequently, 4 Constantly) and an intensity scale (0 Never, 1 not intense to 5 Very Intense). Scores on individual questions are added together to determine a total score. Higher values indicate worse outcomes. The minimum score is 1 and the maximum score is 37.
Distance Visual Acuity | After 1 month of wear
Near Visual Acuity | After 1 month of wear

CONTACTS AND LOCATIONS:
Overall Officials: Jay Mashouf, OD, Principal Investigator — Scripps Optometric Group
Locations (1):
- Scripps Optometric Group, San Diego, California, United States